CLINICAL TRIAL: NCT03685110
Title: Prospective, Non-Interventional, Multicenter, Post-Market Clinical Follow-up Study CoreHip®
Brief Title: CoreHip - Post Market Clinical Follow-Up Study
Status: Active, not recruiting | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1509
Record Dates: First submitted 2018-09-21; First posted 2018-09-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Degenerative Osteoarthritis; Rheumatic Arthritis; Fractures, Hip; Necrosis, Femur Head
Keywords: Hip Arthroplasty; Hip Prosthesis
MeSH Terms: conditions — Joint Diseases; Rheumatic Fever; Hip Fractures; Femur Head Necrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CoreHip: Clinical and Radiological Data of 300 patients of a Standard Patient Population, who are treated with CoreHip Total Hip Arthroplasty for Indications according to the Instructions for Use (IfU) with a five year follow Up
  Interventions: Device: CoreHip Total Hip Arthroplasty

INTERVENTIONS:
Device: CoreHip Total Hip Arthroplasty — Replacement of the Hip Joint

SUMMARY:
The study is designed as a prospective, non-interventional multicentre cohort study. The product under Investigation will be used in Routine clinical practice and according to the authorized Instructions for Use (IfU). Aim of this observational study is to collect clinical and radiological results of the CoreHip® endoprosthesis system in a Standard Patient Population and when used in Routine clinical practice.

DETAILED DESCRIPTION:
The CoreHip® System has a range of different stem designs to address most of the indications and anatomical conditions met in Primary THA patients within one implant and Instrument System.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 18 years
* Indication for THA with a CoreHip® stem
* Written informed consent

Exclusion Criteria:

* Pregnancy
* Patient age < 18 years
* Patient not able to regularly participate at the follow-up examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change of Hip Joint Function measured by Harris Hip Score over time (HHS) | Preoperative, 3 months postoperative, approx. 12-24 months postoperative and approx. 5 years postoperative
  The Harris Hip Score (HHS) assesses the results of hip surgery, evaluates various hip disabilities and methods of treatment in an adult population. The HHS is a clinician-based outcome measure. The domains covered are pain (pain severity and its effect on activities and need for pain medication), function (daily activities (stair use, using public transportation, sitting, and managing shoes and socks) and gait (limp, support needed, and walking distance)), absence of deformity, and range of Motion (hip flexion, adduction, internal rotation, and extremity length discrepancy).
  There are 10 items. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).

SECONDARY OUTCOMES:
Restoration of preoperative leg length | preoperative and 3 months postoperative
  Comparison of preoperative and postoperative leg length
Restoration of preoperative offset | preoperative and 3 months postoperative
  Comparison of preoperative and postoperative Offset angle of the femoral neck
Change of Oxford Hip Score (OHS) over time | Preoperative, 3 months postoperative, approx. 12-24 months postoperative and approx. 5 years postoperative
  A patient-reported outcome instrument which contains 12 questions on activities of daily living that assess function and residual pain in patients undergoing total hip replacement (THR) surgery. The score has a maximum of 48 points (best possible outcome), each question has five answers, ranging from 4 Points (best possible) to 0 Points (worst possible).
Change of Quality of Life (EQ-5D-5L) over time | Preoperative, 3 months postoperative, approx. 12-24 months postoperative and approx. 5 years postoperative
  EuroQol five-dimension scale. A standardised instrument created by the EuroQol Group as a measure of health outcome. EQ-5D is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each of which can take one of five Levels reflecting severity (no problems, slight problems, moderate problems, severe problems and extreme Problems). Each answer results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Change of Radiological results: implant position | Preoperative, 3 months postoperative, approx. 12-24 months postoperative and approx. 5 years postoperative
  Changes in implant Position throughout the follow-up period
Development of Radiological results: radiolucent lines | Preoperative, 3 months postoperative, approx. 12-24 months postoperative and approx. 5 years postoperative
  Development of radiolucent lines ("Gruen" zones) in AP and lateral x-rays throughout the follow-up period
Adverse Events | up to five years
  documentation of all product related adverse Events occuring with the Hip Prosthesis throughout the follow-up period
Survival Rate of the Hip Prosthesis | up to five years
  Survival Analysis of stems in-situ throughout the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Henning Windhagen, Prof. Dr. med., Principal Investigator — Orthopädische Kliniken im Annastift, Medizinische Hochschule Hannover
Locations (6):
- Germany (4):
  - Ortrhopädische Klinik Markgröningen, Markgröningen, Baden-Wurttemberg
  - Orthopädische Chirurgie München, München, Bavaria
  - MHH, Hanover, Lower Saxony
  - St. Josefs Krankenhaus Endoprothetik Zentrum, Salzkotten
- Switzerland (2):
  - Spital Brig, Brig
  - Luzerner Kantonsspital Sursee, Sursee